CLINICAL TRIAL: NCT04261816
Title: Association Between Early Extubation and Postoperative Complications After Liver Transplantation: A Retrospective Propensity Score-matched Analysis
Brief Title: Early Extubation and Postoperative Complications After Liver Transplantation
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Professor, West China Hospital
Other Study IDs: 2020-014
Record Dates: First submitted 2020-02-01; First posted 2020-02-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-04

CONDITIONS: Liver Transplantation
MeSH Terms: interventions — Airway Extubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Operating room extubation group: extubation in the operating room immediately following liver transplantation
  Interventions: Procedure: extubation in the operating room
- ICU extubation group: extubation in the ICU following liver transplantation
  Interventions: Procedure: extubation in the ICU

INTERVENTIONS:
Procedure: extubation in the operating room — Patients who underwent liver transplantation early extubation in the operating room immediately following liver transplantation
  Groups: Operating room extubation group
Procedure: extubation in the ICU — Patients who underwent liver transplantation extubation in the ICU following liver transplantation
  Groups: ICU extubation group

SUMMARY:
This is a retrospective cohort study. Patients who underwent liver transplantation from January 1, 2016 to December 31, 2019 were admitted to the study and divided into two groups. Operating room extubation group: early extubation in the operating room immediately following liver transplantation. Intensive care unit (ICU) extubation group: delay extubation in the ICU following liver transplantation. The primary objectives were to compare the incidence of composite outcome between the two groups. secondary objectives were to compare outcomes such as length of stay, hospital length of stay, and total cost between the two groups.

DETAILED DESCRIPTION:
Patients who underwent liver transplantation from January 1, 2016 to December 31, 2019 were admitted to the study. Inclusion criteria: (1) adult patients (age ≥ 18 years), (2) undergoing liver transplantation. Exclusion criteria were the following: (1) re-transplantation; (2) multi-visceral transplantation; (3) intraoperative death; (4) severe encephalopathy (West Haven criteria III or IV); (5) those who had preoperative mechanical ventilation; (6) incomplete clinical data. The primary objectives was a composite of 30-day all-cause mortality, in-hospital AKI, or in-hospital moderate to severe pulmonary complications. Complications were defined and graded as mild, moderate, or severe as described by European Perioperative Clinical Outcome definitions and were included if they occurred in hospital after surgery. The secondary objectives included in-hospital moderate to severe infectious complications, unplanned reintubation rates, ICU and postoperative hospital lengths of stay, and total hospital cost.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years)
* Undergoing liver transplantation

Exclusion Criteria:

* Re-transplantation
* Multi-organ transplants
* Intra-operative deaths
* severe encephalopathy (West Haven criteria III or IV)
* patients who had preoperative mechanical ventilation or fulminant hepatic failure
* Incomplete clinical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent liver transplantation from January 1, 2016 to December 31, 2019 were admitted to the study.
Sampling Method: Non-Probability Sample
Enrollment: 438 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
The incidence of a composite of 30-day all-cause mortality, AKI and moderate to severe pulmonary complications. | through study completion, an average of 1 year
  Complications were defined and graded as mild, moderate, or severe as described by European Perioperative Clinical Outcome definitions and were included if they occurred in hospital after surgery

SECONDARY OUTCOMES:
The incidence of moderate to severe infectious complications | 30 days
  Complications were defined and graded as mild, moderate, or severe as described by European Perioperative Clinical Outcome definitions and were included if they occurred in hospital after surgery
The incidence of re-intubation. | 30 days
  Reintubation was defined as intubation after extubation of a patient who had been initially tracheal intubated under general anaesthesia
The length of hospital stay | through study completion, an average of 1 year
  Length of hospital stay is the duration of a single episode of hospitalization
The length of ICU stay | through study completion, an average of 1 year
  Length of ICU stay is the duration of a single episode of ICU hospitalization
The total hospital cost | 30 days
  The total hospital cost

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xu Y, Zuo Y, Zhou L, Hao X, Xiao X, Ye M, Bo L, Jiang C, Yang J. Extubation in the operating room results in fewer composite mechanical ventilation-related adverse outcomes in patients after liver transplantation: a retrospective cohort study. BMC Anesthesiol. 2021 Nov 18;21(1):286. doi: 10.1186/s12871-021-01508-1. PMID 34794387